CLINICAL TRIAL: NCT03694184
Title: A Pilot Study of the Effect of Individualized Clinical Management Among Parent/Child Dyads on Continuity of Care and Interaction. Phase 1 : Retrospective Evaluation
Brief Title: A Pilot Study of the Effect of Individualized Clinical Management Among Parent/Child Dyads on Continuity of Care and Interaction
Acronym: Rétro-GUIDANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2017/85
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Child Psychiatry; Psychodynamic Therapy; Continuity/Discontinuity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this project aims to collect retrospective data on the conitinuity/disconitnuity rate for child care in the child psychiatry unit of the université hospital of Besançon, France.

ELIGIBILITY:
Inclusion Criteria:

* Family having with a first consultation request submitted from 2015
* Children aged < 10 years old at the time of the first consultation

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Family having with a first consultation request submitted from 2015 Children aged < 10 years old at the time of the first consultation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
rate of contuinity/discontinuity of child care | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vulliez Lauriane, MD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France